CLINICAL TRIAL: NCT02386800
Title: Open Label, Multi-center, Phase IV Study of Ruxolitinib or Ruxolitinib and Panobinostat Combination, for Patients Who Have Completed Prior Global Novartis or Incyte Sponsored Studies
Brief Title: CINC424A2X01B Rollover Protocol
Status: Active, not recruiting | Phase: Phase 4 | Type: Interventional
Sponsor: Novartis Pharmaceuticals (Industry)
Responsible Party: Sponsor
Organization: Novartis (Industry)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CINC424A2X01B; 2014-003527-22 (EudraCT Number)
Record Dates: First submitted 2015-03-06; First posted 2015-03-12 (Estimated); Last update posted 2025-11-26 (Actual); Status verified 2025-11

CONDITIONS: Primary Myelofibrosis; Polycythemia Vera; Graft Versus Host Disease; Acute Myeloid Leukemia; Thalassemia
Keywords: Myelofibrosis; MF; Polycythemia vera; PV; Acute Graft versus Host Disease; aGvHD; Chronic Graft versus Host Disease; cGvHD; Acute Myeloid Leukemia; AML; Thalassemia; Ruxolitinib; INC424; Panobinostat; LBH589
MeSH Terms: conditions — Primary Myelofibrosis; Polycythemia Vera; Graft vs Host Disease; Leukemia, Myeloid, Acute; Thalassemia; Bronchiolitis Obliterans Syndrome | interventions — ruxolitinib; Panobinostat

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Ruxolitinib monotherapy or ruxolitinib plus panobinostat in combination (Experimental): All participants will receive either ruxolitinib monotherapy or ruxolitinib in combination with panobinostat, at the same dose/schedule that they were taking in the parent study.
  Interventions: Drug: ruxolitinib; Drug: panobinostat

INTERVENTIONS:
Drug: ruxolitinib — ruxolitinib tablets or pediatric oral solution - participants continue ruxolitinib as they received in parent study
  Other Names: INC424; Jakavi
Drug: panobinostat — panobinostat capsules - participants to continue receiving panobinostat in combination with ruxolitinib as per the parent study
  Other Names: LBH589; Farydak

SUMMARY:
This is a long term safety study for patients that have been treated with either ruxolitinib or a combination of ruxolitinib with panobinostat, on a Novartis or Incyte sponsored study, who have been judged by the study Investigator to benefit from ongoing treatment.

DETAILED DESCRIPTION:
This roll-over protocol allows patients from multiple protocols, who are still receiving clinical benefit, to continue their treatment in one study that covers multiple indications. The population for the roll-over study should be consistent with the population defined in the parent studies. The primary eligibility criteria for a patient to enter the roll-over protocol is the participation and completion of a Novartis or Incyte study with ruxolitinib monotherapy or combination of ruxolitinib and panobinostat. Efficacy parameters will not be measured; however safety data and an evaluation of clinical benefit will be collected.

ELIGIBILITY:
Key Inclusion criteria:

1. Patient is currently enrolled in a Novartis GDD or GMA-sponsored or Incyte-sponsored clinical study, are receiving either ruxolitinib or combination of ruxolitinib and panobinostat, and fulfilled all of the requirements of the parent protocol.
2. Patient is currently benefiting from the treatment with ruxolitinib monotherapy or combination of ruxolitinib and panobinostat, as determined by the investigator
3. Patient has demonstrated compliance, as assessed by the investigator, with the parent study protocol requirements
4. Patient currently has no evidence of progressive disease, as determined by the investigator, following previous treatment with ruxolitinib or combination of ruxolitinib and panobinostat

Key Exclusion criteria:

1. Patient has been permanently discontinued from study treatment in the parent study due to any reason.
2. Patient's indication is currently approved and reimbursed in the corresponding country for ruxolitinib monotherapy or combination of ruxolitinib and panobinostat.
3. Pregnant or nursing (lactating) women.
4. Female patients of childbearing potential (e.g. are menstruating) who do not agree to abstinence or, if sexually active, do not agree to the use of highly effective contraception, throughout the study and for up to 30 days after stopping study treatment.

Other protocol-defined Inclusion / Exclusion criteria may apply.

Ages: 1 Month to 100 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 279 (Actual)
Dates: Start 2015-03-05 (Actual); Primary Completion 2027-09-16 (Estimated); Study Completion 2027-09-16 (Estimated)

PRIMARY OUTCOMES:
Incidence and severity of AEs and SAEs | 12 years
  The incidence of treatment-emergent AEs and SAEs (new or worsening from baseline) will be summarized by system organ class and/or preferred term, severity (based on CTCAE grades).

SECONDARY OUTCOMES:
Proportion of participants with clinical benefit as assessed by the investigator at scheduled visits. | 12 years
  The analysis of clinical benefit will be descriptive only and cannot be compared to efficacy results of other studies. In addition, as clinical benefit was only added in protocol amendment 1, it may not be available for all participants.
Incidence and severity of AEs and SAEs by treatment group | 12 years
  AEs and SAEs for participants in the Safety group will be listed and summarized by treatment group (ruxolitinib monotherapy / ruxolitinib + panobinostat combination)

CONTACTS AND LOCATIONS:
Overall Officials: Novartis Pharma, A.G, Study Director — Novartis Pharma, A.G.
Locations (90):
- Australia (9):
  - Novartis Investigative Site, Darlinghurst, New South Wales
  - Novartis Investigative Site, Herston, Queensland
  - Novartis Investigative Site, Wooloongabba, Queensland
  - Novartis Investigative Site, Bedford Park, South Australia
  - Novartis Investigative Site, Box Hill, Victoria
  - Novartis Investigative Site, Clayton, Victoria
  - Novartis Investigative Site, Franston, Victoria
  - Novartis Investigative Site, Perth, Western Australia
  - Novartis Investigative Site, St Leonards
- Belgium (4):
  - Novartis Investigative Site, Leuven, Vlaams Brabant
  - Novartis Investigative Site, Antwerp
  - Novartis Investigative Site, Bruges
  - Novartis Investigative Site, Liège
- Bulgaria (3):
  - Novartis Investigative Site, Pleven
  - Novartis Investigative Site, Plovdiv
  - Novartis Investigative Site, Sofia
- Novartis Investigative Site, Toronto, Ontario, Canada
- Chile (3):
  - Novartis Investigative Site, Viña del Mar, Región de Valparaíso
  - Novartis Investigative Site, Santiago, RM
  - Novartis Investigative Site, Santiago
- China (2):
  - Novartis Investigative Site, Hangzhou, Zhejiang
  - Novartis Investigative Site, Beijing
- Novartis Investigative Site, Paris, France
- Germany (8):
  - Novartis Investigative Site, Dresden, Saxony
  - Novartis Investigative Site, Jena, Thuringia
  - Novartis Investigative Site, Aachen
  - Novartis Investigative Site, Dresden
  - Novartis Investigative Site, Hamburg
  - Novartis Investigative Site, Magdeburg
  - Novartis Investigative Site, Mainz
  - Novartis Investigative Site, Ulm
- Greece (2):
  - Novartis Investigative Site, Athens
  - Novartis Investigative Site, Pátrai
- Hungary (6):
  - Novartis Investigative Site, Debrecen, Hajdu Bihar Megye
  - Novartis Investigative Site, Budapest
  - Novartis Investigative Site, Kaposvár
  - Novartis Investigative Site, Kecskemét
  - Novartis Investigative Site, Szeged
  - Novartis Investigative Site, Szombathely
- Novartis Investigative Site, Pune, Maharashtra, India
- Israel (2):
  - Novartis Investigative Site, Afula
  - Novartis Investigative Site, Jerusalem
- Italy (15):
  - Novartis Investigative Site, Ancona, AN
  - Novartis Investigative Site, Bari, BA
  - Novartis Investigative Site, Bologna, BO
  - Novartis Investigative Site, Brescia, BS
  - Novartis Investigative Site, San Giovanni Rotondo, FG
  - Novartis Investigative Site, Florence, FI
  - Novartis Investigative Site, Milan, MI
  - Novartis Investigative Site, Rozzano, MI
  - Novartis Investigative Site, Palermo, PA
  - Novartis Investigative Site, Pavia, PV
  - Novartis Investigative Site, Reggio Calabria, RC
  - Novartis Investigative Site, Roma, RM
  - Novartis Investigative Site, Orbassano, TO
  - Novartis Investigative Site, Varese, VA
  - Novartis Investigative Site, Napoli
- Japan (7):
  - Novartis Investigative Site, Nagoya, Aichi-ken
  - Novartis Investigative Site, Fukuoka, Fukuoka
  - Novartis Investigative Site, Sapporo, Hokkaido
  - Novartis Investigative Site, Isehara, Kanagawa
  - Novartis Investigative Site, Suita, Osaka
  - Novartis Investigative Site, Bunkyo Ku, Tokyo
  - Novartis Investigative Site, Osaka
- Novartis Investigative Site, Beirut, Lebanon
- Novartis Investigative Site, Monterrey, Nuevo León, Mexico
- Poland (2):
  - Novartis Investigative Site, Gliwice, Silesian Voivodeship
  - Novartis Investigative Site, Wroclaw
- Novartis Investigative Site, Lisbon, Portugal
- Russia (3):
  - Novartis Investigative Site, Moscow
  - Novartis Investigative Site, Petrozavodsk
  - Novartis Investigative Site, Saint Petersburg
- South Africa (4):
  - Novartis Investigative Site, Pretoria, Gauteng
  - Novartis Investigative Site, Soweto, Gauteng
  - Novartis Investigative Site, Cape Town, Western
  - Novartis Investigative Site, Pretoria
- South Korea (2):
  - Novartis Investigative Site, Seoul, Korea
  - Novartis Investigative Site, Seoul
- Spain (3):
  - Novartis Investigative Site, Salamanca, Castille and León
  - Novartis Investigative Site, Barcelona, Catalonia
  - Novartis Investigative Site, Pamplona, Navarre
- Sweden (4):
  - Novartis Investigative Site, Huddinge
  - Novartis Investigative Site, Luleå
  - Novartis Investigative Site, Lund
  - Novartis Investigative Site, Uddevalla
- Novartis Investigative Site, Bangkok, Thailand
- Turkey (Türkiye) (4):
  - Novartis Investigative Site, Istanbul, Fatih
  - Novartis Investigative Site, Kayseri, Melikgazi
  - Novartis Investigative Site, Ankara, Sihhiye-Altindag
  - Novartis Investigative Site, Izmir